CLINICAL TRIAL: NCT07336706
Title: The Effect of Escape Room Simulation on Nursing Students' Knowledge and Academic Self-Efficacy Regarding Stoma Care: A Randomized Controlled Study
Brief Title: The Effect of Escape Room Simulation on Nursing Students' Knowledge and Academic Self-Efficacy Regarding Stoma Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Ankara Yildirim Beyazıt University, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: StomaCareEscapeRoom
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Stoma; ESCAPE ROOM
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All students who agree to participate in the study will be administered the "Descriptive Characteristics Form", the "Stoma Care and Colostomy Irrigation Knowledge Test (pre-test)", and the "Nursing Students Academic Self-Efficacy Scale (pre-test)". Students in the experimental group will be given a lecture on stoma care and irrigation by the researcher. After the training, an escape room simulation will be conducted. Each escape room simulation will be conducted with 6 students, in the form of a pre-information session, an escape room simulation application, and an analysis session. Immediately after the escape room simulation is completed, a debriefing session will be held. After the debriefing session, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.
  Interventions: Other: Escape room simulation
- Control (No Intervention): All students who agree to participate in the study will be administered the "Descriptive Characteristics Form", the "Stoma Care and Colostomy Irrigation Knowledge Test (pre-test)", and the "Nursing Students Academic Self-Efficacy Scale (pre-test)". All students in the control group will receive instruction on stoma care and irrigation using traditional teaching methods provided by the researcher. After the training is completed, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.

INTERVENTIONS:
Other: Escape room simulation — All students who agree to participate in the study will be administered the "Descriptive Characteristics Form", the "Stoma Care and Colostomy Irrigation Knowledge Test (pre-test)", and the "Nursing Students Academic Self-Efficacy Scale (pre-test)". Students in the experimental group will be given a lecture on stoma care and irrigation by the researcher. After the training, an escape room simulation will be conducted. Each escape room simulation will be conducted with 6 students, in the form of a pre-information session, an escape room simulation application, and an analysis session. Immediately after the escape room simulation is completed, a debriefing session will be held. After the debriefing session, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.
  Other Names: Education
  Arms: Intervention

SUMMARY:
This research was planned to determine the effect of escape room simulation on nursing students' knowledge and academic self-efficacy levels regarding stoma care. The research was planned as a randomized controlled trial. This research will be conducted with 60 students of the Nursing Department of Başkent University Faculty of Health Sciences between December 29, 2025 and February 28, 2026. All students who agree to participate in the study will be administered the "Descriptive Characteristics Form", the "Stoma Care and Colostomy Irrigation Knowledge Test (pre-test)", and the "Nursing Students Academic Self-Efficacy Scale (pre-test)". Students will be divided into experimental and control groups using a simple randomization method. Students in the experimental group will be given a lecture on stoma care and irrigation by the researcher. After the training, an escape room simulation will be conducted. Each escape room simulation will be conducted with 6 students, in the form of a pre-information session, an escape room simulation application, and an analysis session. In the pre-information session, the simulation objectives, the purpose of the scenario, the roles within the scenario, and the game rules will be explained, and the escape room and standard patient will be briefly introduced to the students in the meeting room. Then, the students will carry out the scenario and game activity (KAHOOT, Table Game, Card Game, Word Cloud, Crossword Puzzle) with a standard patient in the simulation laboratory prepared as an escape room.

The researcher will act as a facilitator during the escape room simulation application. During the simulation, if the expected steps are not performed correctly or the game activity is not successfully completed, the team has the right to request hints from the facilitator. Immediately after the escape room simulation is completed, a debriefing session will be held. The debriefing session, lasting approximately 20-30 minutes for each team, will take place in the meeting room located directly opposite the escape room. During the debriefing session, students will be encouraged to express their feelings and thoughts, and feedback will be provided by the researcher. After the debriefing session, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.

All students in the control group will receive instruction on stoma care and irrigation using traditional teaching methods provided by the researcher. After the training is completed, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.

Data analysis will be performed using the IBM SPSS Statistics 26 software package.

The main research questions are:

Does escape room simulation increases nursing students' knowledge levels regarding stoma care? Does escape room simulation increases nursing students' academic self-efficacy regarding stoma care?

DETAILED DESCRIPTION:
Stoma is a crucial surgical procedure used to treat digestive or urinary system diseases, facilitating passage for stool and urine, promoting wound healing, and reducing complications. In the US, it is reported that approximately 750,000-1 million people live with stomas, and around 100,000 new stoma surgeries are performed annually. Therefore, nurses assume critical responsibility in stoma care through education, counseling, direct care, and complication management. However, the International Ostomy Guidelines (2020) reveal a lack of knowledge and experience among both clinical nurses and nursing students. Similarly, Zimnicki and Pieper (2018) noted that students have low levels of knowledge and insufficient self-confidence in practicing stoma care. Therefore, it is inevitable that stoma care becomes a fundamental component of the nursing curriculum. Students learn these skills through theoretical training, demonstration methods, and psychomotor skill applications; effective and high-quality training reduces anxiety in clinical practice, increases self-confidence, and facilitates the transition to a professional role. Nurses are responsible for providing safe care by making critical decisions in increasingly complex clinical settings. Therefore, nursing education programs must equip students with the skills to integrate current theoretical knowledge with fundamental practical skills, target behaviors, and professional attitudes. The literature shows that innovative learning methods significantly improve students' exam success and conceptual learning levels compared to traditional approaches; they also strengthen motivation, satisfaction, participation, and interaction. These methods also support self-confidence, communication, and critical thinking skills; and contribute to the more effective application of basic nursing skills by integrating them with theoretical knowledge. Innovative learning methods in nursing education include problem-based learning, collaborative learning, game-based learning, simulation-based learning, case-based learning, web-based learning, and concept maps. Escape room simulations, which combine these methods, have emerged as a remarkable innovation in nursing education in recent years. It has been observed that escape room applications improve students' clinical decision-making, communication, teamwork, and problem-solving skills, and studies on this topic are rapidly increasing in the literature. No studies have been found in the literature examining the application of escape room simulation for stoma care on nursing students. Therefore, it is predicted that escape room simulation will increase nursing students' knowledge levels and academic self-efficacy regarding stoma care.

This research was planned to determine the effect of escape room simulation on nursing students' knowledge and academic self-efficacy levels regarding stoma care.

Materials and Methods Study Design The research was planned as a randomized controlled trial with a pre-test-post-test-follow-up design with experimental and control groups.

Research Hypotheses H1: Escape room simulation increases nursing students' knowledge levels regarding stoma care.

H2: Escape room simulation increases nursing students' academic self-efficacy regarding stoma care.

Study Location and Characteristics This research will be conducted with students of the Nursing Department of Başkent University Faculty of Health Sciences between December 29, 2025 and February 28, 2026. The research will be implemented in the Professional Skills Laboratory of Başkent University Faculty of Health Sciences.

Research Population and Sample The research population will consist of 85 students studying in the third year of the Nursing Department of Başkent University Faculty of Health Sciences between December 29, 2025 and February 28, 2026. The research sample will consist of students who meet the inclusion criteria and those who do not meet the exclusion criteria.

Inclusion criteria for the study:

* Being an undergraduate nursing student
* Voluntarily agreeing to participate in the study

Exclusion criteria for the study:

* Being a graduate of any health sciences department
* Having experience with escape room simulation

Data to be excluded:

• Students who do not complete the research process for any reason will be excluded from the study.

The topic of stoma care and irrigation is taught theoretically for two hours in the second year within the scope of the Differentiation and Care in Health Status 1 course. The theoretical content of the courses is explained by faculty members and stoma and wound care nurses using lecture, question-and-answer, and discussion methods.

Randomized Students will be divided into experimental and control groups using a simple randomization method according to their average stoma care knowledge score. Power analysis was performed to calculate the sample size of the study. The G-Power 3.1.9.7 statistical program was used to calculate the sample size of the study. In the study conducted by Aktaş (2023), the effect size related to the difference in knowledge and skill level was determined as 0.903. In the G-Power statistical program, a 5% margin of error, an effect size of 0.903, and a power level of 90% were used. The power analysis determined that the study should be conducted with at least 54 students in total, with 27 students in the experimental group and 27 in the control group. Considering data loss, the sample size was increased by 10%, aiming to reach 60 students.

Data Collection Tools The research data will be collected using the "Descriptive Characteristics Form", the "Stoma Care and Colostomy Irrigation Knowledge Test", and the "Nursing Students Academic General Self-Efficacy Scale".

Descriptive Characteristics Form, this form was prepared by the researchers. The form consists of 5 questions regarding the students' descriptive characteristics (age, gender, general grade point average, etc.) Stoma Care and Colostomy Irrigation Knowledge Test (pre-test-post-test), The Stoma Care and Colostomy Irrigation Knowledge Test, developed and validated by Kulakaç and Çilingir (2024), determines students' knowledge of stoma care and colostomy irrigation. In the form consisting of four-option multiple-choice questions, students' correct answers were evaluated as one point and incorrect answers as zero points. The Stoma Care and Colostomy Irrigation Knowledge Test contains 20 questions on the subject, and the lowest score is zero (0) and the highest is 20. Higher scores indicate higher achievement.

Nursing Students Academic Self-Efficacy Scale (ANSEs), Bulfone et al. Developed by (2019) to determine the academic self-efficacy of nursing students studying at the undergraduate level, and validated and validated in Turkish by Aktay and Çiçek Korkmaz (2023), the scale consists of 14 items and four sub-dimensions. The scale comprises the following sub-dimensions: internal emotion management (items 1, 2, 3), self-control behavior (items 4, 5, 6, 7), external emotion management (items 8, 9, 10, 11), and sociability (items 12, 13, 14). The item scores range from 1 to 5, and the question "How much confidence do you have in yourself?" is scored using a 5-point Likert scale (1 = I have no confidence in myself, 5 = I have a lot of confidence in myself). As the scores obtained from the scale increase, the academic self-efficacy of nursing students increases. There are no items in the scale that are reverse-scored. The Cronbach alpha value of the original scale is 0.84, while in this study it is 0.82.

Data Collection All students who agree to participate in the study will be administered the "Descriptive Characteristics Form", the "Stoma Care and Colostomy Irrigation Knowledge Test (pre-test)", and the "Nursing Students Academic Self-Efficacy Scale (pre-test)". Students will be divided into experimental and control groups using a simple randomization method. Students in the experimental group will be given a lecture on stoma care and irrigation by the researcher. After the training, an escape room simulation will be conducted. Each escape room simulation will be conducted with 6 students, in the form of a pre-information session, an escape room simulation application, and an analysis session. In the pre-information session, the simulation objectives, the purpose of the scenario, the roles within the scenario, and the game rules will be explained, and the escape room and standard patient will be briefly introduced to the students in the meeting room. Then, the students will carry out the scenario and game activity (KAHOOT, Table Game, Card Game, Word Cloud, Crossword Puzzle) with a standard patient in the simulation laboratory prepared as an escape room.

The researcher will act as a facilitator during the escape room simulation application. During the simulation, if the expected steps are not performed correctly or the game activity is not successfully completed, the team has the right to request hints from the facilitator. Immediately after the escape room simulation is completed, a debriefing session will be held. The debriefing session, lasting approximately 20-30 minutes for each team, will take place in the meeting room located directly opposite the escape room. During the debriefing session, students will be encouraged to express their feelings and thoughts, and feedback will be provided by the researcher. After the debriefing session, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.

All students in the control group will receive instruction on stoma care and irrigation using traditional teaching methods provided by the researcher. After the training is completed, and after 1 month the "Stoma Care and Colostomy Irrigation Knowledge Test (post-test)" and the "Nursing Students Academic Self-Efficacy Scale (post-test)" will be administered.

Data Evaluation Data analysis will be performed using the IBM SPSS Statistics 26 software package. When evaluating the study data, frequencies (number, percentage) will be given for categorical variables, and descriptive statistics (mean, standard deviation, median, minimum, maximum) will be given for numerical variables. The Shapiro-Wilk Normality Test will be performed to check the normality assumptions of numerical variables. Differences between two independent groups will be checked using the Mann-Whitney U test, and differences between two dependent numerical variables will be checked using the Wilcoxon analysis. Relationships between two independent numerical variables will be interpreted using Spearman's Rho Correlation Coefficient. Statistical significance will be interpreted at the 0.05 level in the analyses.

Ethical Principles and Permissions Permission obtained from the Başkent University Faculty of Social and Human Sciences Ethics Committee. Permission will be obtained from the Dean's Office of the Faculty of Health Sciences for the implementation of the research. Students participating in the study will be informed face-to-face about the purpose, methodology, potential benefits and risks, voluntary participation principles, and confidentiality policies of the research. Following this, students will be provided with written consent, and each student who provides signed consent will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate nursing student
* Voluntarily agreeing to participate in the study

Exclusion Criteria:

* Being a graduate of any health sciences department
* Having experience with escape room simulation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Stoma Care and Colostomy Irrigation Knowledge Test (pretest-posttest) | Day 1 (pre-education), Day 1 (post-education) and Day 30 (post-education)
  The Stoma Care and Colostomy Irrigation Knowledge Test, developed and validated by Kulakaç and Çilingir (2024), determines students' knowledge of stoma care and colostomy irrigation. In the form consisting of four-option multiple-choice questions, students' correct answers were evaluated as one point and incorrect answers as zero points. The Stoma Care and Colostomy Irrigation Knowledge Test contains 20 questions on the subject, and the lowest score is zero (0) and the highest is 20. Higher scores indicate higher achievement.
Nursing Students Academic Self-Efficacy Scale | Day 1 (pre-education), Day 1 (post-education) and Day 30 (post-education)
  Bulfone et al. developed by (2019) to determine the academic self-efficacy of nursing students studying at the undergraduate level, and validated and validated in Turkish by Aktay and Çiçek Korkmaz (2023), the scale consists of 14 items and four sub-dimensions. The scale comprises the following sub-dimensions: internal emotion management (items 1, 2, 3), self-control behavior (items 4, 5, 6, 7), external emotion management (items 8, 9, 10, 11), and sociability (items 12, 13, 14). The item scores range from 1 to 5, and the question "How much confidence do you have in yourself?" is scored using a 5-point Likert scale (1 = I have no confidence in myself, 5 = I have a lot of confidence in myself). As the scores obtained from the scale increase, the academic self-efficacy of nursing students increases. There are no items in the scale that are reverse-scored. The Cronbach alpha value of the original scale is 0.84, while in this study it is 0.82.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)